CLINICAL TRIAL: NCT05220345
Title: Synergistic Effect of G-Eye Balloon for Behind the Folds Visualization With Artificial Intelligence Assisted Polyp Detection (Discovery System) on Adenoma Detection Rate. 'Discovery III Study'
Brief Title: Synergistic Effect of G-Eye Balloon for Behind the Folds Visualization With CADe (Discovery System) on Adenoma Detection Rate.
Acronym: DiscoveryIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: PENTAX Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL80004.091.21
Record Dates: First submitted 2022-01-31; First posted 2022-02-02 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Polyp; Colonoscopy; Artificial Intelligence; Adenoma
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Intervention Model Description: International multicenter prospective interventional cohort, compared with a cohort from the Discovery II study (NL73127.091.20, trial code NL9135).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- colonoscopy with a combined BFT and CADe assisted approach (Other): This multicenter single-arm colonoscopy trial will compare colonoscopy assisted by both balloon-BFT visualizing and CADe to CADe-only assisted colonoscopy in diagnostic, screening (non-iFOBT based)), or surveillance colonoscopy. The latter group will be selected from the interventional arm from the Discovery II trial, using corresponding participating centers. All subjects in this trial will undergo the same treatment, i.e., combined balloon and CADe-assisted colonoscopy.
  Interventions: Device: colonoscopy assisted by both balloon-Behind The Folds visualizing and Computer assisted detection (CADe)

INTERVENTIONS:
Device: colonoscopy assisted by both balloon-Behind The Folds visualizing and Computer assisted detection (CADe) — All participants will be subjected to a colonoscopy procedure, assisted by both G-eye balloon and the Discovery CADe system. Standard of care regarding the colonoscopy procedure will be applied to all study subjects. Any lesions detected during the procedure will be removed directly

SUMMARY:
Colonoscopy is the gold standard for colorectal screening. The diagnostic accuracy of colonoscopy highly depends on the quality of inspection of the colon during the procedure. To increase detection new polyp detection systems based on artificial intelligence (AI) have been developed. However, these systems still depend on the ability of the endoscopist to adequately visualize the complete colonic mucosa, especially to detect smaller and more subtle lesions, or lesions hidden behind folds in the colon. With this study we want to combine a device to flatten the folds in the colon combined with an artificial intelligence system to further improve the detection rate of lesions during colonoscopy.

DETAILED DESCRIPTION:
Rationale: Colonoscopy is the gold standard for CRC screening. The adenoma detection rate (ADR) is the most important quality parameter for colonoscopy, because of its inverse association with the risk of interval CRC. Yet, the adenoma miss rate (AMR) in conventional colonoscopy is reported in meta-analyses to vary between 22-26%. The diagnostic accuracy of colonoscopy highly depends on the quality of inspection of the colonic mucosa during the procedure. To increase the adenoma detection rate (ADR), new polyp/adenoma detection systems based on artificial intelligence (AI) have been developed, i.e., computer assisted detection (CADe). However, these systems still depend on the ability of the endoscopist to adequately visualize the complete colonic mucosa, especially to detect smaller and more subtle lesions. Therefore, we hypothesize that ADR can further be improved by combining a CADe system, the Discovery system, with a behind the fold (BTF) visualization technique, the G-Eye.

Study design: International multicenter prospective interventional cohort, compared with a cohort from the Discovery II study (NL73127.091.20, trial code NL9135). All subjects will be undergoing colonoscopy with a combined BFT and CADe assisted approach. Outcomes will be corrected for confounders using regression modeling.

Study population: 194 Adult patients (>18 years) from 3 hospitals, scheduled for diagnostic, screening (non-iFOBT based), or surveillance colonoscopy. Exclusion criteria: inflammatory bowel disease (IBD), known polyp or tumor upon referral, therapeutic procedure (e.g. endoscopic mucosal resection), prior surgical resection of any portion of the colon, American Society of Anesthesiologists score of ≥3, Inadequately corrected anticoagulation disorders or anticoagulation medication use, inability to provide informed consent.

Main study endpoints: The primary objective of the present study is to compare ADR between CADe assisted and a combined BTF/CADe assisted colonoscopy. Secondary objectives include advanced neoplasia rate (including advanced adenomas and/or CRC), polyp detection rate, size and histopathology, mean number of polyps per patient, procedure times, bowel cleaning levels, adverse events, inter-operator variability.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Eligible patients who are scheduled for surveillance colonoscopy will undergo one BFT and CADe assisted colonoscopy. There will be no burden for participants regarding the colonoscopy procedure. Colonoscopy is a commonly performed procedure, and the overall serious adverse event rate is low with an estimated risk 2.8 per 1000 colonoscopies. The risk of experiencing a (serious) adverse event with G-Eye and Discovery guided colonoscopy is believed to be equivalent to conventional colonoscopy. The benefit for patients is a higher likelihood of lesion detection during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Referred and scheduled for diagnostic, screening (non-iFOBT based), or surveillance colonoscopy.

Exclusion Criteria:

* Inflammatory bowel disease (IBD)
* Known polyp or tumor upon referral
* Therapeutic procedure (e.g., endoscopic mucosal resection)
* Prior surgical resection of any portion of the colon
* American Society of Anesthesiologists score of ≥3
* Inadequately corrected anticoagulation disorder or anticoagulation medication use
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | 30 days after procedure
  Calculated as the number of patients in whom at least one adenoma is detected during the colonoscopy procedure, divided by the total number of patients that underwent the colonoscopy procedure.

SECONDARY OUTCOMES:
Advanced adenoma detection rate (AADR). | 30 days after procedure
  calculated as the number of patients in whom at least one advanced adenoma is detected during the colonoscopy procedure, divided by the total number of patients that underwent the colonoscopy procedure
Polyp Detection Rate | 30 days after procedure
  calculated as the number of patients in whom at least one polyp is detected during the colonoscopy procedure, divided by the total number of patients that underwent the colonoscopy procedure
Sessile detection Rate | 30 days after procedure
  calculated as the number of patients in whom at least one SSL is detected during the colonoscopy procedure, divided by the total number of patients that underwent the colonoscopy procedure
Indication specific ADR, | 30 days after procedure
  ADR specific for screening, diagnostic, or surveillance
Mean number of adenomas detected per patient | 30 days after procedure
  Mean number of adenomas detected per patient
Mean number of polyps detected per patient | 30 days after procedure
  Mean number of polyps detected per patient
Number of sessile serrated lesions | 30 days after procedure
  Number of sessile serrated lesions
Number of advanced adenomas (adenomas ≥ 10 mm and/or with a villous component and/or with HGD | 30 days after procedure
  Number of advanced adenomas (adenomas ≥ 10 mm and/or with a villous component and/or with HGD
Size of the lesion subdivided in categories 0-5 mm, 6-10 mm, 10-20 mm, >20 mm | During procedure
  Size of the lesion subdivided in categories 0-5 mm, 6-10 mm, 10-20 mm, >20 mm
Location of the lesion: cecum, ascending colon, transverse colon, descending colon, sigmoid, rectum; | During procedure
  Location of the lesion: cecum, ascending colon, transverse colon, descending colon, sigmoid, rectum;
Morphological characteristics of the lesion using the Paris classification (Ip, Is, IIa, IIb, IIc, III) | During procedure
  Morphological characteristics of the lesion using the Paris classification (Ip, Is, IIa, IIb, IIc, III)
Histopathological characteristics of the lesion according to the Vienna classification | 30 days after procedure
  Histopathological characteristics of the lesion according to the Vienna classification
ADR of the first 20% of patients that have undergone colonoscopy by each endoscopist will be compared with the final 20% of patients in each arm to identify any changes in ADR throughout the trial | At end of study
  ADR of the first 20% of patients that have undergone colonoscopy by each endoscopist will be compared with the final 20% of patients in each arm to identify any changes in ADR throughout the trial
Bowel cleansing | During procedure
  Using the Boston Bowel Prep Scale
Cecal intubation rate (CIR) | During procedure
  Cecal intubation rate (CIR)
Procedure times with both techniques (i.e., total procedure time, mean polypectomy time and withdrawal time) | During procedure
  Procedure times with both techniques (i.e., total procedure time, mean polypectomy time and withdrawal time)
Severe) adverse events (S)AEs up to 30 days post-procedure | 30 days after procedure
  SAEs will be subcategorized into colonoscopy related, cardiac (cardiac ischemia, heart failure, arrhythmia, other) pulmonary (exacerbation COPD, infectious, other), neurological (stroke, cerebrovascular accident, bleeding, other), and other (surgical interventions etc.)
Gloucester Comfort Scale score and analgesia use | During procedure
  Gloucester Comfort Scale score and analgesia use
Post-colonoscopy surveillance intervals when applying European and US surveillance guidelines | 30 days after procedure
  Post-colonoscopy surveillance intervals when applying European and US surveillance guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Siersema, Prof, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center Nijmegen, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The dataset used during this study is available from the corresponding author upon reasonable request.